CLINICAL TRIAL: NCT06279481
Title: Effect of Virtual Reality (VR) on Pain Relieve During Colonoscopy: A Prospective Randomized Controlled Study
Brief Title: Effect of Virtual Reality (VR) on Pain Relieve During Colonoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-K2458
Record Dates: First submitted 2023-12-22; First posted 2024-02-28 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-02

CONDITIONS: Pain; Colonoscopy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: a single-centered, prospective, randomized controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The virtual reality hardware includes a headset (OLED display mode), a headset cable, a High-Definition Multimedia (HDM) cable, a processor unit, an Alternating Current (AC) power converter, a six-axis dynamic sensing system (three-axis gyroscope, three-axis accelerator sensor), a cinema AC screen, and a camera. The software that patients would be engaged in is highly interactive and requires total attention for about 15 minutes. The device would be tried out by the patients prior to the operation.
  Interventions: Other: Nonpharmacological method
- Control (No Intervention): Patients undergo traditional colonoscopy procedures.

INTERVENTIONS:
Other: Nonpharmacological method — Virtual reality
  Arms: Virtual Reality

SUMMARY:
Purpose: To evaluate the effectiveness and safety of virtual reality (VR) technology in alleviating pain during colonoscopy.

Design and Methods: In the context of a single-centered, prospective, randomized controlled study, the pain levels experienced during colonoscopy are compared between the VR group and the control group.

DETAILED DESCRIPTION:
Patient allocation to either the VR group or the control group will be determined through a randomization process employing sealed opaque envelopes. Patients in the VR group will engage in interactive gaming experiences facilitated by VR devices. The primary outcome measure will be the assessment of pain levels during colonoscopy, which will be quantified using the "Visual Analogue Scale." Additionally, researchers will assess anxiety levels using the "State-Trait Anxiety Inventory" both before and after the colonoscopy procedure. Vital signs during colonoscopy, procedural effects, and adverse effects would also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age
* Able to cooperate and complete the questionnaires independently
* Stable vital signs with no serious cardiovascular or cerebrovascular diseases
* Voluntary participation

Exclusion Criteria:

* Severely impaired in vision or hearing to accommodate VR devices
* Previous history of anxiety, depression, cognitive impairment, balance disorder, mental illness, or epilepsy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of Visual Analogue Scale Mean Scores by Groups | Evaluated immediately after colonoscopy.
  Pain scoring will apply the Visual Analogue Scale (VAS), which is a visual measurement using an axis rated by 0-10, with 0 for painless and 10 for the severest pain. Subjects will report the lightest score, average score, and highest score regarding pain during colonoscopy, and the mean score will be calculated. The emotional change caused by pain and attention given to the presence of pain will also be reported to adjust the main outcome.

SECONDARY OUTCOMES:
Comparison of State Trait Anxiety Inventory Mean Scores by Groups | Evaluated immediately both prior and after colonoscopy.
  State Trait Anxiety Inventory evaluates anxiety with a scale containing 20 items, scoring between 20 points (no anxiety) to 80 points (high anxiety).
Comparison of Vital Signs between Groups: Pulse Rate | Evaluated both before and every 3 minutes during colonoscopy.
  All vital signs of patients will be measured by a same multifunctional ECG monitor.
Comparison of Vital Signs between Groups: Blood Pressure | Evaluated both before and every 3 minutes during colonoscopy.
  All vital signs of patients will be measured by a same multifunctional ECG monitor.
Comparison of Vital Signs between Groups: Respiration Rate | Evaluated both before and every 3 minutes during colonoscopy.
  All vital signs of patients will be measured by a same multifunctional ECG monitor.
Comparison of Vital Signs between Groups: Oxygen Saturation | Evaluated both before and every 3 minutes during colonoscopy.
  All vital signs of patients will be measured by a same multifunctional ECG monitor.
Comparison of Patient Satisfaction of Colonoscopy between Groups | Evaluated immediately after colonoscopy.
  Patient satisfaction will be assessed by a self-made rating form. Results will be reported on a scale of 1-5 with a higher score standing for higher satisfaction. Results will be adjusted by bowel preparation, cecal intubation rate, and procedural duration.
Comparison of Patient Willingness of Future Colonoscopy between Groups | Evaluated immediately after colonoscopy.
  Patient willingness to undergo future colonoscopies will be assessed by a self-made rating form. Results will be reported on a scale of 1-5 with a higher score standing for higher willingness. Results will be adjusted by bowel preparation, cecal intubation rate, and procedural duration.
Comparison of Adverse Effects in both groups | During and immediately after colonoscopy.
  Any adverse effect (e.g. nausea, vomiting, headache, or dizziness) would be immediately recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yingyun Yang, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No